CLINICAL TRIAL: NCT03778099
Title: The Effect of Cinnamon on Ovulation Induction in Women With Polycystic Ovary Syndrome, Jeddah 2019: Randomized Double-blind Placebo-controlled Trial
Brief Title: The Effect of Cinnamon on Ovulation Induction in Women With Polycystic Ovary Syndrome
Acronym: PCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr. Wael Alzhrani, Principle Investigator, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W-001
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Polycystic Ovary Syndrome; Ovulation
Keywords: PCOS; Ovulation; Cinnamon
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon Group (Experimental): Two capsules of cinnamon 500mg twice per day after meals (2g/day). All capsules will be given simultaneously with the clomiphene citrate medication (standard treatment for infertility in women with PCOS). Participants will be asked to keep their normal lifestyle including daily food and physical activity level.
  Interventions: Drug: Cinnamon Cap 500 MG
- Placebo Group (Placebo Comparator): Placebo capsules will contain 450 mg of starch and 50 mg of cinnamon powder (to improve blindness regarding taste and odor). Color, shape, and size of placebo capsules will be exactly the same as the cinnamon capsules.
  2g/day along with clomiphene citrate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinnamon Cap 500 MG — The Cinnamomum cassia (C. aromaticum) capsules will be purchase from Spring Valley company (distributed by Wal-Mart Stores, Inc. USA) by the investigator.
  Arms: Cinnamon Group
Drug: Placebo — 450 mg of starch and 50 mg of cinnamon powder
  Arms: Placebo Group

SUMMARY:
Title: The effect of cinnamon supplementation on ovulation induction in women with polycystic ovary syndrome, Jeddah 2019: Randomized Double-Blind Placebo-controlled trial

Phase: III

Population: 118 women with polycystic ovary syndrome will be recruited from Obstetrics and Gynecology clinics in King Abdul-Aziz University Hospital, Jeddah 2019.

Subject Participation Duration: Each participant will be followed for three months.

Intervention: 2g of cinnamon capsules daily will be provided.

Objectives:

Primary Objective:

1. To compare the effectiveness of cinnamon supplement in combination with clomiphene citrate versus clomiphene citrate alone on ovulation in women with PCOS, in King Abdul-Aziz University Hospital in Jeddah 2019.
2. To measure the difference in insulin resistance after three months of cinnamon supplementation in women with PCOS in King Abdul-Aziz University Hospital, Jeddah 2019.
3. To determine the effect of cinnamon and CC on menstrual cyclicity, approximated by menstrual frequency, during the study period, in women with PCOS in King Abdul-Aziz University Hospital, Jeddah 2019
4. To evaluate the quality of life in women with PCOS in King Abdul-Aziz University Hospital, Jeddah 2019.

Secondary Objectives:

* To measure the pregnancy rate in women with PCOS in King Abdul-Aziz University Hospital, Jeddah 2019

Description of Study Design:

The participants will be randomized in 1:1 fashion. Allocation concealment will be ensured using similar bottles labeled by letters A and B, to receive either the combination of cinnamon supplement and clomiphene citrate or clomiphene citrate with placebo.

First visit: Patients will be evaluated during the early follicular phase for progesterone level and HOMA-IR and QUICK-I. Follow up: 3 months.

Last Visit: Patients will be re-evaluated to compare the difference.

ELIGIBILITY:
Inclusion Criteria:

* Married women aged 18-40 seeking to become pregnant, meeting the Rotterdam criteria for polycystic ovary syndrome

Exclusion Criteria:

* Current pregnancy or lactation.
* Current use of treatment of infertility.
* Established diagnosis of diabetes mellitus.
* Use of Insulin-sensitizing treatment within the past three months.
* Hormonal treatment involving estrogen or progesterone within the past three months.
* Known hypersensitivity to cinnamon.
* Use of statin medication.
* Any other supplements that contain cinnamon within the past month.
* BMI <18.5 or BMI >35.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with PCOS
Enrollment: 33 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Ovulation Confirmation by Progesterone level | 3 months
  Progesterone level > 3ng/mL or pregnancy confirmed
Changes in insulin resistance | 3 months
  HOMA-IR
Menstrual frequency | 3 months
  No. of menses/ No. of months
Quality of life: Infertility quality of life questionnaire | 6 months
  The 36 FertiQoL items are rated according to 5 types of response scales.
  The response scales are:
  Very poor (0), poor (1), neither poor nor good (2), very good (4) Very dissatisfied (0), dissatisfied (1), neither satisfied nor dissatisfied (2), satisfied (3), very satisfied (4) Always (0), very often (1), quite often (2), Seldom (3), never (4) An extreme amount (0), very much (1), a moderate amount (2), a little (3), not at all (4) Completely (0), a great deal (1), moderately (2), not much (3), not at all (4)
  Scores on the response scales are reversed, summed and scaled to range from 0 to 100. Higher scores on the subscales and total scores indicate better quality of life.

SECONDARY OUTCOMES:
Pregnancy Rate | 3 months
  Number of pregnancies including live births, induced abortions, and fetal deaths / Number of women aged 18 - 40 years) × 1,000

CONTACTS AND LOCATIONS:
Overall Officials: Wael H Alzhrani, Principal Investigator
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided